CLINICAL TRIAL: NCT02229435
Title: Laboratory Database-based Analysis of the Interdisciplinary Urologic-nephrological Care of the Chronic Kidney Disease (CKD) With Estimated Glomerular Filtration Rate (eGFR) Under 60 ml/Min of the Population in Saxony-Anhalt / Metropolitan Area Magdeburg.
Brief Title: Urologic-nephrological Care of Chronic Kidney Disease in Saxony-Anhalt/Magdeburg.
Acronym: UroCKDisS
Status: Completed | Type: Observational
Sponsor: University of Magdeburg (Other)
Collaborators: Medical Laboratory Schenk-Ansorge Magdeburg Germany. (Unknown)
Responsible Party: Principal Investigator, Johann J. Wendler, MD, Dr. med., University of Magdeburg
Other Study IDs: URO-MD-040
Record Dates: First submitted 2014-08-26; First posted 2014-09-01 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Chronic Kidney Disease (CKD)
Keywords: Chronic kidney disease; Urological care; Nephrological care
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- eGFR <60ml/min: Patients with CKD with eGFR <60 ml/min (CKD-EPI or MDRD) 12/2004-08/2014 of Medical Laboratory, Prof. Schenk / Dr. Ansorge and Colleagues, GbR, Am Neustädter Feld 47, 39124 Magdeburg, Germany.

SUMMARY:
Statement:

Patients with Chronic kidney disease (CKD) with an estimated glomerular filtration rate (eGFR) under 60 ml/min using the MDRD-6 (Modification of Diet in Renal Disease) formula and/or CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) formula should undergo nephrological and urological care (diagnosis and treatment) to prevent chronic kidney failure. This is recommended by the National Kidney Foundation Kidney Disease Outcomes Quality Initiative (KDOQI), Kidney Disease Improving Global Outcomes (KDIGO) and European Urological Association (EAU). Renal and postrenal diseases can cause or worsen CKD. Internistic and intrarenal diseases can caused or worsen CKD. All diseases affecting CKD should be treated and the medical care should be optimized.

Hypothesis:

Not all patients with CKD receive urological and nephrological care. Interdisciplinary work of outpatient working urologists and nephrologists in the metropolitan area Magdeburg / Saxony-Anhalt Germany is unknown. An descriptive analysis of interdisciplinary treatment connection of CKD patients for an orientating statement is needed.

DETAILED DESCRIPTION:
The Medical Laboratory Schenk-Ansorge Magdeburg Saxony-Anhalt Germany receives all blood samples of outpatient patients of the medical practices of the metropolitan area Magdeburg Saxony-Anhalt Germany. Every patient has a lifetime identification number Independent of the submitting practice. Every submitting medical doctor has a lifetime identification number and is identified by her/his medical subject /specialization. This analysis is based on that laboratory database. For that study a cohort of 1.031.336 patients from 12/2004 to 08/2014 is evaluated, that had been received blood tests with measurement of serum creatinine. For every serum creatinine an eGGR is calculated with the guideline recommended formula.

ELIGIBILITY:
Inclusion Criteria:

* Measured serum creatinine and estimated glomerular filtration rate
* eGFR < 60 ml/min

Exclusion Criteria:

* dialysis
* no serum creatinine measured
* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All sampled outpatient patients (blood tests with measurement of serum creatinine) 12/2004-08/2014 of the medical laboratory Prof. Schenk / Dr. Ansorge and Colleagues, GbR, Am Neustädter Feld 47, 39124 Magdeburg, metroplitan area Magdeburg Saxony-Anhalt, Germany.
Sampling Method: Non-Probability Sample
Enrollment: 1031336 (Actual)
Dates: Start 2004-12; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Chronic kidney disease | 1 year
  % of outpatient patients with eGFR < 60 ml/min and interdisciplinary urological and nephrological care in metropolitan area Magdeburg, Saxony-Anhalt, Germany.

CONTACTS AND LOCATIONS:
Overall Officials: Johann J Wendler, Dr., Principal Investigator — Urology University Magdeburg; Martin Schostak, Prof. Dr., Study Chair — Urology University Magdeburg; Herwart Schenk, Prof. Dr., Study Director — Medical Laboratory Am Neustädter Feld 47, 39124 Magdeburg, Saxony-Anhalt, Germany.; Constanze Tienken, Cand. med., Principal Investigator — Doctorand Urology University Magdeburg
Locations (1):
- Department of Urology University Magdeburg, Magdeburg, Saxony-Anhalt, Germany

REFERENCES:
- See also: Medical Laboratory Schenk-Ansorge Magdeburg, Germany. — http://www.schenk-ansorge.de/Kontakt.aspx
- See also: Department of Urology University Magdeburg, Germany. — http://urologie.uni-magdeburg.de/urologie.html